CLINICAL TRIAL: NCT01070706
Title: Phase Ib/II Study of Primary Chemotherapy With Paclitaxel, Gemcitabine, and Sunitinib in Patients With HER2-negative Stage II/III Breast Cancer
Brief Title: Phase Ib/II Study of Primary Chemotherapy With Paclitaxel, Gemcitabine, and Sunitinib
Acronym: PGS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jungsil Ro (Other Government)
Collaborators: Pfizer (Industry); HK inno.N Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jungsil Ro, Chief, Center for Clinical Trials, National Cancer Center, Korea, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-08-369
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Patients with HER2- stage II/III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel, Gemcitabine, Sunitinib (Experimental): Paclitaxel, Gemcitabine, Sunitinib
  Interventions: Drug: Paclitaxel,Gemcitabine,Sunitinib

INTERVENTIONS:
Drug: Paclitaxel,Gemcitabine,Sunitinib — To determine the MTD, only DLT occurring during the first cycle of treatment will be considered. And MTD is defined as the dose level at which at least one-third of patients experience a DLT during their first treatment course. The recommended dose level for the subsequent phase II study is defined as the preceding dose level before the MTD is attained.
  If MTD is not reached, the recommended initial dose of the phase II part will be at the dose of paclitaxel 80 mg/m2 and gemcitabine 1200 mg/m2 (days 1, 8) with sunitinib 37.5 mg qd D2-D15.
  Other Names: PGS

SUMMARY:
Phase Ib part:

▪ Primary objective: To demonstrate the recommended dose of the combination of paclitaxel, gemcitabine, and sunitinib (sutene®) (PGS) as preoperative chemotherapy in patients with HER2-negative operable breast cancer

* Secondary objective:

  1. To demonstrate the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of this regimen
  2. To determine the safety profile

     Phase II part
* Primary objective:

To evaluate the pathologic complete response rate (pCR) to preoperative administration of PGS

▪ Secondary objective:

1. To assess breast conserving rate after preoperative PGS
2. To evaluate clinical response rate, disease free survival (DFS), and overall survival (OS)
3. To assess the safety profiles of PGS

DETAILED DESCRIPTION:
Unlike adjuvant chemotherapy, primary (preoperative) chemotherapy will shrink tumor and allow more patients to become candidates for conservative surgery and avoid mastectomy. It also is an in vivo chemosensitivity test and the result is a predictive marker for clinical outcomes.

Paclitaxel has been shown to be an effective agent in the treatment of breast cancer. Gemcitabine is a cytosine arabinoside prodrug analog and shows response rates of 15% to 46% as a single agent with very low toxicity. The combination of paclitaxel and gemcitabine (PG) resulted in improvement in objective response rate, time to progression and overall survival compared to paclitaxel monotherapy in patients with metastatic breast cancer. In addition, primary chemotherapies with PG and PGH (PG + trastuzumab) showed significant activity and very low toxicity in phase II studies performed at National Cancer Center, Korea (ASCO 2007 and SABCS 2008, respectively).

Sunitinib is an oral small molecular tyrosine kinase inhibitor that exhibits potent anti-angiogenic and antitumor activity. Sunitinib is a rationally designed small molecule that inhibits members of the split-kinase domain family of receptor tyrosine kinases (RTKs) including the vascular endothelial growth factors (VEGFs) types 1, 2, and 3, platelet-derived growth factor receptor (PDGFR)-α, and -β, stem cell factor receptor (KIT), colony stimulating factor 1 receptor (CSF-1R), Fms-like tyrosine kinase (FLT-3), and glial cell line-derived neurotrophic factor receptor (RET). Inhibition of these RTKs blocks signal transduction, thereby affecting many of the process involved in tumor growth, progression, metastasis, and angiogenesis. Angiogenesis plays a vital role in the growth and metastasis of solid tumors. Preclinical and indirect clinical evidence has accumulated to support the role of neo-angiogenesis in the pathogenesis and progression of breast cancer. Breast cancer neo-vascularization, as measured by an increase in microvessel density, is correlated with the extent of disease and is associated with vascular invasion of the tumor, a prerequisite for blood-borne metastasis. VEGFR signaling is also implicated in the pathobiology of breast cancer. Breast cancer patients exhibit high levels of circulating VEGF and other RTKs are very likely implicated in breast cancer pathogenesis.

Interestingly, a phase II study (Study A6181002) of single-agent sunitinib (50 mg/d on schedule 4/2) in breast cancer patients with anthracycline- and taxane-refractory metastatic disease revealed a response rate of approximately 14% in 51 assessable patients, leading to additional accrual.

When sunitinib is combined with paclitaxel, significant activity was noticed with tolerable toxicity profile in a phase I trial (SABCS 2007). Based on this trial, phase III trial of paclitaxel and sunitinib is ongoing. In addition, phase I trials of gemcitabine and sunitinib combination are ongoing.

Based both on the significant activity of PG combination regimens in the neoadjuvant and metastatic setting and on the phase I trials of combination regimens with sunitinib-paclitaxel and sunitinib-gemcitabine, we plan to conduct a phase IB/II study of primary chemotherapy with sunitinib, paclitaxel and gemcitabine in patients with HER2-negative stage II/III breast cancer. The goal of this phase IB/II study is to define the recommended dose and maximum tolerable dose of paclitaxel and gemcitabine in combination with sunitinib, and explore the activity of this combination as preoperative chemotherapy in patients with HER2-negative operable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. ECOG performance status 0-2
3. Histologically confirmed and newly diagnosed breast cancer
4. Documented HER2/neu non-overexpressing or non-amplified disease

   * 0-1+ by HER2 IHC or
   * HER2 gene non-amplification by HER2 FISH
5. Clinical stage II or III operable breast cancer
6. Axillary node positivity determined by cytology
7. No prior hormonal, chemotherapy or radiotherapy is allowed
8. No breast operation other than biopsy to make diagnosis is allowed
9. Adequate hematologic, hepatic and renal function

   * Absolute neutrophil count ≥ 1,500/μL
   * Hemoglobin ≥ 10.0 g/dL
   * Platelet ≥ 100,000/μL
   * AST/ALT ≤ 2 X UNL (upper limit of normal)
   * Total bilirubin ≤ 1.5 mg/dL
   * Alkaline phosphatase ≤ 2 X UNL
   * Serum creatinine ≤ 1.5 mg/dL
10. Adequate cardiac function LVEF ≥ 50% and within the institutional range of normal as measured by echocardiogram or MUGA scan within 4 weeks of enrollment
11. Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to registration
12. Normal mental function to understand and sign the consent

Exclusion Criteria:

1. Patients with metastatic breast cancer
2. Patients who received hormonal, chemotherapy or radiotherapy for breast cancer
3. Patients who underwent surgery for breast cancer
4. Patients with T2N0, or inflammatory (T4d) breast cancer
5. Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer
6. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
7. Any of the following within the 12 months prior to starting study treatment

   * severe, unstable angina
   * Myocardial infarction
   * Uncontrolled or symptomatic congestive heart failure
   * coronary/peripheral artery bypass graft
   * cerebrovascular accident including transient ischemic attack
   * pulmonary embolism
8. Ongoing cardiac dysrhythmias of grade ≥2, atrial fibrillation of any grade, or QTc interval >470 msec.
9. Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy)
10. Current treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg po daily for deep vein thrombosis prophylaxis is allowed).
11. Known HIV infection
12. Pregnancy or breastfeeding. Female patients who are pregnant or nursing, female of child-bearing potential who is unwilling to use adequate contraception to prevent pregnancy during the program. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to study entry.
13. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug during administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Phase Ib part: To demonstrate the recommended dose of the combination of paclitaxel, gemcitabine, and sunitinib. Phase II part: To evaluate the pathologic complete response rate (pCR) | 17Mar2009~08Apr2010

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, Principal Investigator — Chief, Center for Breast Cancer, National Cancer Center, Korea
Locations (1):
- Center for breast cancer, National Cancer Center, Goyang, Kyeonggido, South Korea